CLINICAL TRIAL: NCT04101461
Title: The Effectiveness of Single Versus Double Daily Dose of Oral Iron on the Prevention of Iron Deficiency Anemia in Obese Pregnant Women
Brief Title: The Oral Iron on the Prevention of Iron Deficiency Anemia in Obese Pregnant
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Lecturer, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IDA-Obese
Record Dates: First submitted 2019-09-22; First posted 2019-09-24 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Anemia of Pregnancy
MeSH Terms: interventions — Iron; Blood Cell Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I: 27 mg elemental iron (Active Comparator): will receive PharaFerro27; Devart Lab Company, Egypt; once daily starting at 12 -14 weeks until 37-38 weeks
  Interventions: Drug: Iron; Diagnostic Test: Complete blood count; Diagnostic Test: Serum ferritin; Diagnostic Test: Serum hepcidin; Diagnostic Test: Serum Iron; Diagnostic Test: Serum total iron binding capacity
- Group II: 54 mg elemental iron (Active Comparator): will receive two tablets of PharaFerro27; Devart Lab Company, Egypt; daily starting at 12 -14 weeks until 37-38 weeks
  Interventions: Drug: Iron; Diagnostic Test: Complete blood count; Diagnostic Test: Serum ferritin; Diagnostic Test: Serum hepcidin; Diagnostic Test: Serum Iron; Diagnostic Test: Serum total iron binding capacity

INTERVENTIONS:
Drug: Iron — PharaFerro27; Devart Lab Company, Egypt
Diagnostic Test: Complete blood count — to assess the anemia
Diagnostic Test: Serum ferritin — to assess the anemia
Diagnostic Test: Serum hepcidin — to assess the iron abosrption
Diagnostic Test: Serum Iron — to assess the anemia
Diagnostic Test: Serum total iron binding capacity — to assess the anemia

SUMMARY:
Anemia is known as a condition in which the hemoglobin level is lower than normal. Anemia is one of the most common complications during pregnancy. Anemia in pregnancy is defined as a hemoglobin level < 110 g/L . Anemia is an important risk factor in pregnancy which leads to both maternal and fetal morbidity and mortality.

The pregnant woman needs more iron during pregnancy, so iron deficiency anemia is very common during pregnancy. In Egypt; iron deficiency anemia affects about one in every two pregnant women, especially in rural areas. Pregnant women require about 27 mg/day elemental iron to cover their increased need. The pregnant women should start taking a daily supplement of 30mg of elemental iron as a preventive measure against iron deficiency anemia especially in poor countries.

Obesity is defined as having an excessive amount of body fat. The body mass index, a measurement based on height and weight, determines the obese if the figure more than 30 kg/m2. There is an increased rate of overweight and obesity among pregnant women. According to the World Health Organization, 46% of adult females in Egypt are obese.

Many researches in the literature revealed a strong relationship between high BMI in pregnancy and iron deficiency anemia. Hepcidin is an iron regulating hormone in the body. Increases in iron levels in the plasma stimulate the production of hepcidin, which blocks iron absorption from the diet, so; hepcidin production is suppressed in the case of iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant woman in a singleton pregnancy (12-14 weeks).
2. BMI (30- 40 kg/m2).
3. Normal hemoglobin level (>11 g/dL).
4. Normal hematocrit (Hct 31-41%).
5. Normal ferritin level (6-130 ng/mL).
6. Women willingness to participate in the study.
7. Women living in the nearby area to make follow-up visits possible.

Exclusion Criteria:

1. Multiple gestations.
2. Women received a recent blood transfusion.
3. Women with threatened miscarriage.
4. Women are known to have pathological blood loss.
5. Intolerant to oral iron form.
6. History of the hematologic disorder.
7. Women used iron in the past 3 months.
8. Women with chronic diseases (hypertension, diabetes, renal diseases, thyroid disease……).

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 230 (Actual)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
The number of anemic women at time of delivery | 6 months

SECONDARY OUTCOMES:
The mean level of maternal Hemoglobin at 37-38 weeks . | 6 months
The incidence of patients' reported side effect | 6 months
The difference in serum ferritin | 6 months
The difference in serum hepcidin | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Woman's Health Hospital - Assiut university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided